CLINICAL TRIAL: NCT06907368
Title: Analysis of the Functional Impact of Total Knee Arthroplasty Using Quantified Gait Analysis and Proprioceptive Evaluation. Prospective, Single-center, Open-label Study, Cohort Follow-up.
Brief Title: Analysis of the Functional Impact of Total Knee Arthroplasty Using Quantified Gait Analysis and Proprioceptive Evaluation
Acronym: ARTHROPROMA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0425
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Total Knee Arthroplasty for Gonarthrosis
Keywords: Gonarthrosis; Proprioception; Functional recovery; Patient-reported Outcomes Measures (PROMs); Quantitative Gait Analysis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quantitative Gait Analysis — The following explorations will be carried out pre-operatively (pre-OP), then post-operatively at 3 months (post-OP3) and 12 months (post-OP12) :
  * Quantified gait analysis (QGA)
  * Functional tests (mechanical analysis of everyday tasks):
    * SIT-TO-STAND test (test consisting of standing up and sitting down on a chair)
    * STEP INITIATION test (test consisting of walking up a step and then down)
  * Proprioceptive tests :
    * Joint Position Sense (JPS) (angle memorization and reproduction test at the knee joint)
    * OBSTACLE CLEARANCE test (test consisting in simulating the clearance of an obstacle)
  * Questionnaires :
    * Functional questionnaires :
    * KSS (Knee Society Score)
    * SKV (Simple knee value)
    * KOOS (Knee Injury and Osteoarthritis Outcome Score)
    * Quality of life (EQ5D-5L) The total duration of each exploration session is estimated at 1 hour .
  Other Names: Functional tests; Proprioceptive tests; Questionnaires

SUMMARY:
Total knee arthroplasty remains the gold standard in the management of disabling gonarthrosis. Improved functional results, increased availability of care and an ageing population have all contributed to the rise in total knee replacement surgery in Western countries. Surgical techniques have been steadily improving for several decades in terms of implant positioning and joint alignment. However, 10% of patients are dissatisfied with the clinical and functional results. The challenge is to understand why these patients remain dissatisfied despite these surgical advances. Our aim is to understand the functional impact of knee prosthesis through a quantified analysis of gait, the performance of certain tasks of daily living, and pre- and post-operative proprioceptive assessments. We will link these results with patient feedback to identify factors potentially responsible for poor postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Gonarthrosis on imaging with indication for total knee arthroplasty (TKA)
* Isolated gonarthrosis

Exclusion Criteria:

* Patient objecting to study participation
* Patient with an associated pathology causing balance and/or proprioceptive disorders (Parkinson's, stroke sequelae, etc.).
* Patients with a history of cognitive disorders, either confirmed or currently being assessed.
* IADL score below 3, indicating major dependence in daily life.
* Patients unable to walk without technical aids for 6 months.
* Patients unable to get up from a chair without armrests
* Parker score below 6
* Protected persons covered by articles L1121-5 to L1121-8 of the French Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who undergone total knee arthroplasty for gonarthrosis in Grenoble University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative functional recovery of patients who have undergone total knee arthroplasty for gonarthrosis by analyzing their locomotion ability | Preoperatively (PreOP) and 12 months postoperatively (PostOP12)
  The primary endpoint is a composite endpoint assessed by quantified gait analysis (QGA) :
  1/ Gait speed 2 / Step length

SECONDARY OUTCOMES:
Functional recovery by analyzing changes in gait variability | Preoperatively (PreOP) , 3 months postoperatively (PostOP3), 12 months postoperatively (PostOP3)
  Functional recovery is assessed by quantified gait analysis (QGA) :
  Measurement of step length Measurement of step width Measurement of cycle time Measurement of step speed and cadence Measurement of gait variability and stability parameters
Impact of total knee arthroplasty (TKA) on proprioception | Preoperatively (PreOP) , 3 months postoperatively (PostOP3), 12 months postoperatively (PostOP3)
  Proprioception is assessed by Joint Position Sense (JPS) test :
  Error between target angle and established angle: average absolute error in relation to the target angle in degrees. This will enable us to obtain an average absolute error for the three trials for each target angle per lower limb and per patient.
Functional recovery after TKA by analyzing changes in daily living tasks by SIT TO STAND test | Preoperatively (PreOP) , 3 months postoperatively (PostOP3), 12 months postoperatively (PostOP3)
  Measurement of displacements of the center of pressure and gravity, angular velocities (trunk, knee, hip, ankle), hip and knee angular moments, ground reaction force (for each lower limb).
Functional recovery after TKA by analyzing changes in daily living tasks by STEP INITIATION test | Preoperatively (PreOP) , 3 months postoperatively (PostOP3), 12 months postoperatively (PostOP3)
  Analysis of ground reaction force on healthy side vs. pathological side during ascent and descent of step, knee joint amplitudes in flexion during ascent and descent of step.
Functional recovery after TKA by analyzing changes in daily living tasks by OBSTACLE CLEARANCE test | Preoperatively (PreOP) , 3 months postoperatively (PostOP3), 12 months postoperatively (PostOP3)
  * Analysis of obstacle-crossing accuracy (minimum foot-to-obstacle distance and distance covered by the lower limb, taking the center of the ankle as reference, until the obstacle is crossed).
  * Analysis of variability: Variability in the position of the center of the ankle when passing the obstacle + variability in the trajectory of the lower limb (hip and knee angles + angular velocity of the hip and knee).
  * Analysis of movement symmetry: Symmetry between the legs, based on the vertical distance foot-obstacle during clearance, and on the similarity index based on angles and angular velocity of the hip, knee and trunk.
Evolution of Quality of Life | Preoperatively (PreOP) , 3 months postoperatively (PostOP3), 12 months postoperatively (PostOP3)
  EQ5D-5L questionnaire
Evolution of the patient's functional results assessed by the KSS questionnaire | Preoperatively (PreOP) , 3 months postoperatively (PostOP3), 12 months postoperatively (PostOP3)
  The KSS is a functional questionnaire (e.g. questions on pain, joint amplitude, possible walking distance) completed by the patient and the surgeon.
Evolution of the patient's functional results assessed by the SKV questionnaire | Preoperatively (PreOP) , 3 months postoperatively (PostOP3), 12 months postoperatively (PostOP3)
  The SKV score is a very simple functional score, based on a single question: "How would you rate your knee on the day of the examination, compared with a normal knee in percentage terms?" completed by the patient.
Evolution of the patient's functional results assessed by the KOOS questionnaire | Preoperatively (PreOP) , 3 months postoperatively (PostOP3), 12 months postoperatively (PostOP3)
  KOOS is a questionnaire assessing knee function, pain and impact on daily life score to be completed exclusively by the patient. The questionnaire comprises five dimensions: symptoms, stiffness, pain, function of daily life and activities, sports and leisure.

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided